CLINICAL TRIAL: NCT00858871
Title: A Randomized, Double-blind, Multi-center Phase III Study of Brivanib Versus Sorafenib as First-line Treatment in Patients With Advanced Hepatocellular Carcinoma
Brief Title: First Line Hepato Cellular Carcinoma (HCC)
Acronym: BRISK FL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA182-033; EUDRACT # 2008-003533-24
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Hepato Cellular Carcinoma (HCC)
MeSH Terms: interventions — brivanib; Sorafenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brivanib (Active Comparator)
  Interventions: Drug: Brivanib; Drug: Placebo
- Sorafenib (Active Comparator)
  Interventions: Drug: Sorafenib; Drug: Placebo

INTERVENTIONS:
Drug: Brivanib — Tablets, Oral, 800 mg, Once Daily, Until disease progression or unacceptable toxicity
  Other Names: BMS-582664
  Arms: Brivanib
Drug: Placebo — Capsules, Oral, twice Daily, Until disease progression or unacceptable toxicity
  Arms: Brivanib
Drug: Sorafenib — Capsules, Oral, 800 mg, twice daily, Until disease progression or unacceptable toxicity
  Arms: Sorafenib
Drug: Placebo — Tablets, Oral, Once Daily, Until disease progression or unacceptable toxicity
  Arms: Sorafenib

SUMMARY:
The purpose of this study is to compare the overall survival of brivanib versus sorafenib in subjects with advanced HCC who have not received prior systemic therapy.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Histologic or cytologic confirmed diagnosis of HCC.
* Advanced HCC: disease not eligible for surgical and/or locoregional therapies OR progressive disease after surgical and/or locoregional therapies
* Child-Pugh Class A
* ECOG performance status 0-1
* Adequate hematologic, hepatic, and renal function

Exclusion Criteria:

* Prior use of any systemic anti-cancer chemotherapy, immunotherapy or molecular targeted agents for HCC
* History of active cardiac disease
* Thrombotic or embolic events within the past 6 months (except HCC tumor thrombus)
* Any other hemorrhage/bleeding event >= CTCAE Grade 3 within 8 weeks except for esophageal or gastric varices
* Inability to swallow tablets or untreated malabsorption syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1714 (Actual)
Dates: Start 2009-05; Primary Completion 2012-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
To compare the overall survival of brivanib versus sorafenib in subjects with advanced HCC who have not received prior systemic treatment | Survival will be assessed continuously

SECONDARY OUTCOMES:
To compare the time to progression (TTP) (investigator assessed using modified RECIST criteria for HCC | Every 6 weeks
To compare the investigator assessed objective response rate (ORR) and disease control rate (DCR) using modified RECIST criteria for HCC | Every 6 weeks
To determine duration of response, duration of disease control, and time to response (TTR) | Every 6 weeks
To assess the safety profile of brivanib and sorafenib | Every 6 weeks
To explore PK and exposure-response in the study population | Every 6 weeks
To compare time to symptomatic progression | Every 6 weeks
To compare health-related quality of life | Every 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (146):
- United States (12):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Univ Of Ark For Med Sci, Little Rock, Arkansas
  - Agajanian Institute Of Hematology And Oncology, Downey, California
  - Sharp Clinical Oncology Research, San Diego, California
  - Va Ct Healthcare System, West Haven, Connecticut
  - Medical Specialists Of Palm Beaches, Lake Worth, Florida
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - 3912 Taubman Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Thomas Jefferson Univ., Philadelphia, Pennsylvania
  - Mcguire Dvamc, Richmond, Virginia
  - University Of Wisconsin, Madison, Wisconsin
- Argentina (4):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Caba, Buenos Aires
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, Rosario, Santa Fe Province
- Australia (5):
  - Local Institution, Camperdown, New South Wales
  - Local Institution, Concord, New South Wales
  - Local Institution, Westmead Nsw, New South Wales
  - Local Institution, Parkville, Victoria
  - Local Institution, Prahan, Victoria
- Local Institution, Liège, Belgium
- Brazil (10):
  - Local Institution, Fortaleza, Ceará
  - Local Institution, Salvador, Estado de Bahia
  - Local Institution, Salvador - Ba, Estado de Bahia
  - Local Institution, Goiânia, Goiás
  - Local Institution, Divinópolis, Minas Gerais
  - Local Institution, Curitiba, Paraná
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Barretos, São Paulo
  - Local Institution, Jaú, São Paulo
  - Local Institution, São Paulo, São Paulo
- Canada (4):
  - Local Institution, Calgary, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, London, Ontario
  - Local Institution, Montreal, Quebec
- China (15):
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Chongqing, Chongqing Municipality
  - Local Institution, Guangzhou, Guangdong
  - Local Institution, Guanzhou, Guangdong
  - Local Institution, Nanning, Guangxi
  - Local Institution, Wuhan, Hubei
  - Local Institution, Changsha, Hunan
  - Local Institution, Changzhou, Jiangsu
  - Local Institution, Nanjing, Jiangsu
  - Local Institution, Suzhou, Jiangsu
  - Local Institution, Dalian, Liaoning
  - Local Institution, Xi'an, Shaanxi
  - Local Institution, Shanghai, Shanghai Municipality
  - Local Institution, Chengdu, Sichuan
  - Local Institution, Hangzhou, Zhejiang
- Czechia (2):
  - Local Institution, Brno
  - Local Institution, Prague
- France (10):
  - Local Institution, Bordeaux
  - Local Institution, Clichy
  - Local Institution, Créteil
  - Local Institution, Grenoble
  - Local Institution, Lille
  - Local Institution, Lyon
  - Local Institution, Marseille
  - Local Institution, Paris
  - Local Institution, Rennes
  - Local Institution, Vandœuvre-lès-Nancy
- Germany (5):
  - Local Institution, Berlin
  - Local Institution, Halle
  - Local Institution, Hamburg
  - Local Institution, Magdeburg
  - Local Institution, Ulm
- Hong Kong (2):
  - Local Institution, Hong Kong
  - Local Institution, Shatin
- India (11):
  - Local Institution, Hyderabad, Andhra Pradesh
  - Local Institution, Kochi, Kerala
  - Local Institution, Trivandrum, Kerala
  - Local Institution, Pune, Maharashtra
  - Local Institution, Ahmedabad
  - Local Institution, Chennai
  - Local Institution, Coimbatore
  - Local Institution, Hyderabad
  - Local Institution, Kolkata
  - Local Institution, Mumbai
  - Local Institution, New Delhi
- Italy (5):
  - Local Institution, Milan
  - Local Institution, Napoli
  - Local Institution, Pisa
  - Local Institution, Roma
  - Local Institution, Torrette -Ancona
- Japan (16):
  - Local Institution, Kashiwa-shi, Chiba
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Kanazawa, Ishikawa-ken
  - Local Institution, Kawasaki-shi, Kanagawa
  - Local Institution, Yokohama, Kanagawa
  - Local Institution, Tsu, Mie-ken
  - Local Institution, Okayama, Okayama-ken
  - Local Institution, Higashinari-ku, Osaka
  - Local Institution, Osaka, Osaka
  - Local Institution, Ōsaka-sayama, Osaka
  - Local Institution, Sunto-gun, Shizuoka
  - Local Institution, Chuo-Ku, Tokyo
  - Local Institution, Minato-ku, Tokyo
  - Local Institution, Musashino-shi, Tokyo
  - Local Institution, Shimonoseki-shi, Yamaguchi
  - Local Institution, Nishinomiya-shi
- Mexico (6):
  - Local Institution, Aguascalientes, Aguascalientes
  - Local Institution, D.f., Mexico City
  - Local Institution, Distrito Federal, Mexico City
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Tlalpan, Mexico City
  - Local Institution, Monterrey, Nuevo León
- Poland (4):
  - Local Institution, Gdansk
  - Local Institution, Gliwice
  - Local Institution, Krakow
  - Local Institution, Warsaw
- Local Institution, San Juan, Pr, Puerto Rico
- Local Institution, Moscow, Russia
- South Africa (5):
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Durban, KwaZulu-Natal
  - Local Institution, Cape Town, Western Cape
  - Local Institution, Observatory, Cape Town, Western Cape
  - Local Institution, Rondebosch, Western Cape
- South Korea (5):
  - Local Institution, Busan
  - Local Institution, Daegu
  - Local Institution, Gyeonggi-do
  - Local Institution, Kyunggi-do
  - Local Institution, Seoul
- Spain (3):
  - Local Institution, Santiago de Compostela, A Coruna
  - Local Institution, Alicante
  - Local Institution, Barcelona
- Sweden (2):
  - Local Institution, Stockholm
  - Local Institution, Uppsala
- Taiwan (6):
  - Local Institution, Changhua
  - Local Institution, Kaohsiung City
  - Local Institution, Taichung
  - Local Institution, Tainan R.o.c.
  - Local Institution, Taipei
  - Local Institution, Taoyuan District
- Local Institution, Bangkok, Thailand
- Turkey (Türkiye) (5):
  - Local Institution, Ankara
  - Local Institution, Antalya
  - Local Institution, Istanbul
  - Local Institution, Izmir
  - Local Institution, Kayseri
- United Kingdom (5):
  - Local Institution, Bristol, Avon
  - Local Institution, London, Greater London
  - Local Institution, Manchester, Greater Manchester
  - Local Institution, Birmingham, West Midlands
  - Local Institution, Leeds, Yorkshire

REFERENCES:
- [Derived] Kolamunnage-Dona R, Berhane S, Potts H, Williams EH, Tanner J, Janowitz T, Hoare M, Johnson P. Sorafenib is associated with a reduced rate of tumour growth and liver function deterioration in HCV-induced hepatocellular carcinoma. J Hepatol. 2021 Oct;75(4):879-887. doi: 10.1016/j.jhep.2021.05.015. Epub 2021 May 27. PMID 34052255
- [Derived] Johnson PJ, Qin S, Park JW, Poon RT, Raoul JL, Philip PA, Hsu CH, Hu TH, Heo J, Xu J, Lu L, Chao Y, Boucher E, Han KH, Paik SW, Robles-Avina J, Kudo M, Yan L, Sobhonslidsuk A, Komov D, Decaens T, Tak WY, Jeng LB, Liu D, Ezzeddine R, Walters I, Cheng AL. Brivanib versus sorafenib as first-line therapy in patients with unresectable, advanced hepatocellular carcinoma: results from the randomized phase III BRISK-FL study. J Clin Oncol. 2013 Oct 1;31(28):3517-24. doi: 10.1200/JCO.2012.48.4410. Epub 2013 Aug 26. PMID 23980084
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx